CLINICAL TRIAL: NCT00140816
Title: Dairy Products and Metabolic Effects - A Multicentre Nordic Study
Brief Title: Dairy Products and Metabolic Effects (Norwegian Part)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Tine (Industry); Opplysningskontoret for meieriprodukter. (Unknown); The Research Council of Norway (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Melk61015
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-02

CONDITIONS: Metabolic Syndrome X; Heart Disease
MeSH Terms: conditions — Metabolic Syndrome; Heart Diseases

INTERVENTIONS:
Behavioral: Increased intake of dairy products

SUMMARY:
Foods containing more dairy fat (and thus a higher proportion of short and medium chain fatty acids and possibly some other nutrients or micronutrients with effect on energy intake, satiety or energy metabolism) affect energy balance and metabolic profile in subjects prone to develop abdominal adiposity and metabolic syndrome.

The aim of the study is to test the hypothesis that intake of dairy products has a favorable effect on markers of the metabolic syndrome.

To explore such a hypothesis the participants have to be in a free living situation during an extended study period.

ELIGIBILITY:
Inclusion Criteria:

Apparently healthy men and women aged 30-65 years with:

* BMI < 35 kg/m2.
* Having signed a written informed consent
* Limited habitual intake of dairy products according to dietary questionnaire.
* Traits of the metabolic syndrome - two or more of the following criteria fulfilled:

  * Fasting plasma glucose ≥ 6.1 mmol/l
  * Serum triglycerides ≥ 1.7 mmol/l
  * Serum HDL cholesterol < 1.0 mmol/l (40 mg/dl) (men) and < 1.3 mmol/l (50 mg/dl) (women)
  * Blood pressure ≥130/ 85 mmHg
  * Waist circumference >94cm (men) and >88cm (women).

Exclusion Criteria:

Patients with any of the following conditions will not be included in the trial:

* Known Type 1 diabetes, or treated type 2 diabetes.
* With HbA1c ≥ 7,5% at the first blood sample.
* Pregnant or lactating women.
* Known abnormal thyroid hormone levels, or high thyroid stimulating hormone (TSH) level.
* Having received an investigational drug in the last 30 days before date of randomisation.
* Unable or unwilling to comply with the protocol.
* Likely to withdraw from the study before its completion.

Concomitant medications:

* With a lipid lowering drug (fibrate, statin) within the last 6 weeks before randomisation.
* Treated with antidiabetic drugs.
* Treated with Cyclosporin A.
* Change within the last 6 weeks before randomisation and during the study in the medications that could interfere with the lipid profile (i.e., anti- hypertensive drugs, oral corticosteroids, thyroid hormones, retinoids, thiazidic derivative, hormone replacement therapy).
* Treated with oral anticoagulants.
* Treated with protease inhibitors (indinavir, ritonavir, saquinavir)
* Treated against obesity: medical treatment within the last 6 weeks (orlistat, sibutramine) and/or surgery (gastroplasty, bypass).

Associated diseases or conditions:

* Diabetic ketoacidosis, diabetic pre-coma.
* Current chronic pancreatitis, or identified risk or known history of acute pancreatitis.
* Hepatic insufficiency, acute alcohol intoxication, alcoholism.
* Known cholelithiasis without cholecystectomy.
* AST and/or ALT > 2 times the upper normal limit (UNL).
* Renal failure or renal dysfunction defined by serum creatinine levels > 135 µmol/L in males and > 110 µmol/L in females.
* Recent myocardial infarction (within 3 months prior to randomisation),
* Known gastric or peptic ulcer or intestinal disease within the previous 3 months of randomisation capable of modifying the intestinal absorption of the drugs.
* Any other severe pathology such as cancer, mental illness, etc, which in the opinion of the investigator might pose a risk to the patient or confound the results of the study.
* Blood pressure >160/100 mmHg.
* Body weight changes exceeding ± 5% of total body weight during the last three months before admission. Drugs affecting lipid and glucose metabolism, weight reducing drugs, antihypertensives and other drugs with known metabolic effects.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Weight
Body mass index (BMI)
Waist circumference/sagittal abdominal diameter
Proportion of body fat (bioelectrical impedance analysis [BIA], dual energy x-ray absorptiometry [DEXA])
Serum lipids (triglycerides [TG], cholesterol [chol], high-density lipoprotein [HDL] chol, low-density lipoprotein [LDL] chol, apolipoprotein (apo) B, apo A1, fatty acid composition)
Blood glucose, HbA1c%
Serum insulin, C-peptide
Blood pressure (systolic blood pressure [SBP], diastolic blood pressure [DBP])
Marker of fibrinolysis: plasminogen activator inhibitor [PAI-1]
Markers for inflammation: micro C-reactive protein (microCRP), interleukin-6 (IL-6), 15-keto-DH-prostaglandin F2 alfa (in urine), fibrinogen
Markers of endothelial function: vascular cell adhesion molecule (VCAM), vWillebrand factor
Lipid peroxidation ("oxidative stress"): 8-F2-isoprostanes (in urine)

SECONDARY OUTCOMES:
Adiponectin, leptin
LDL particle size
Gene expression in leukocytes
Direct measurement of insulin sensitivity
Glucose tolerance test (0, 30, 60, 90, 120)
Fat load test (0, 4, 6)
Serum free fatty acids (FFA)
Fat content of faeces
Polymorphisms in genes with direct influence on relation between endogen lipid synthesis and lipid oxidation (AMP-kinase, SREBP1c, stearoyl desaturase-SCD1, acetyl-CoA carboxylase-ACC2, acyl-CoA synthetase-ACS1)

CONTACTS AND LOCATIONS:
Overall Officials: Jan I Pedersen, Prof. dr. med., Principal Investigator — Inst. of Basic Medical Sciences, Dept. of Nutrition, University of Oslo
Locations (1):
- Lipidklinikken, Medisinsk avdeling, Rikshospitalet, Oslo, Norway